CLINICAL TRIAL: NCT05656456
Title: The Impact of the COVID-19 Pandemic on Patients With Obsessive-Compulsive Disorder and Their live-in Family Members
Brief Title: Impact of COVID-19 on Mental Health of OCD Patients and live-in Family Members
Acronym: COVIDOCS
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-07561
Record Dates: First submitted 2022-12-15; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Family accommodation; Covid-19
MeSH Terms: conditions — Obsessive-Compulsive Disorder; COVID-19 | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OCD patients: Patients with obsessive-compulsive disorder
  Interventions: Other: Y-BOCS or FAS online survey, interview
- live-in family members: Live-in family members of OCD patients
  Interventions: Other: Y-BOCS or FAS online survey, interview

INTERVENTIONS:
Other: Y-BOCS or FAS online survey, interview — Y-BOCS or FAS and online survey will be administered interview will be conducted

SUMMARY:
The impact of the current Covid-19 pandemic on mental health of people with preexisting psychiatric problems is enormous. This longitudinal study investigates the prevalence of mental health problems (obsessive compulsive, or depressive symptoms, anxiety, stress...) of obsessive-compulsive disorder (OCD) patients and their live-in family members. We also aim to investigate the impact of the pandemic, isolation measures, exposure to media and changing therapeutic setting in OCD patients and their live-in family members through qualitative research.

DETAILED DESCRIPTION:
The impact of the current Covid-19 pandemic on mental health of people with preexisting psychiatric problems is enormous. Previous studies during the SARS outbreak demonstrated a significant burden and increase of mental health problems in people with preexisting psychiatric problems, but little is known about the impact on preexisting obsessive-compulsive disorder (OCD). This longitudinal study aims to investigate the prevalence of mental health problems of OCD patients during and after the Covid-19 pandemic. We also want to investigate the impact on family accommodation (FA). There is growing evidence that FA maintains and/or facilitates OCD symptoms. OCD patients and their live-in family members, followed at the Centre for OCD of the Ghent university hospital, will be included. Sociodemographic data, data regarding employment and previous mental health problems will be collected at the first survey. The Y-BOCS (OCD symtoms) and FAS (family accommodation) will be taken from patients and family members respectively at the start, after 1, 3 and 6 months. The Depression, Anxiety and Stress Scale (DASS-21), the Dutch translation of the Covid-19 Peritraumatic Distress Index (CPDI) will be administered at the same time points through an online survey.

Secondly, patients and live-in family members will be interviewed about their experiences concerning the covid pandemic, the isolation measures, media exposure and change of mental health practice and the impact on the OCD (qualitative research).

ELIGIBILITY:
Inclusion Criteria:

* OCD patients
* live-in family members of OCD patients

Exclusion Criteria:

* not speaking fluently Dutch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: OCD patients followed at the Centre of OCD and their live-in family members
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2020-11-22 (Actual); Study Completion 2020-11-22 (Actual)

PRIMARY OUTCOMES:
OCD symptoms in patients at baseline | Baseline
  OCD symptoms as measured by the Y-BOCS
Family accommodation in family members at baseline | Baseline
  FA as measured by the family accommodation scale (FAS)
Change in OCD symptoms in patients | Baseline + 30 days, baseline + 90 days, baseline + 180 days
  OCD symptoms as measured by the Y-BOCS
Change in family accommodation in family members | Baseline + 30 days, baseline + 90 days, baseline + 180 days
  FA as measured by the family accommodation scale (FAS)

SECONDARY OUTCOMES:
Depressive symptoms at baseline in patients and family members | Baseline
  Depressive symptoms as measured by the 7-item depression subscale of the self-reported 21-item Depression, Anxiety, and Stress Scale (DASS-21) (DASS-21-Depression). A higher score indicates more depressive symptoms with a minimum score of 0 and a maximum score of 21.
Change in depressive symptoms in patients and family members | Baseline + 30 days, baseline + 90 days, baseline + 180 days
  Depressive symptoms as measured by the 7-item depression subscale of the self-reported 21-item Depression, Anxiety, and Stress Scale (DASS-21) (DASS-21-Depression). A higher score indicates more depressive symptoms with a minimum score of 0 and a maximum score of 21.
Anxiety symptoms at baseline in patients and family members | Baseline
  Anxiety symptoms as measured by the 7-item depression subscale of the self-reported 21-item Depression, Anxiety, and Stress Scale (DASS-21) (DASS-21-Depression). A higher score indicates more anxiety symptoms with a minimum score of 0 and a maximum score of 21.
Change in anxiety symptoms in patients and family members | Baseline + 30 days, baseline + 90 days, baseline + 180 days
  Anxiety symptoms as measured by the 7-item depression subscale of the self-reported 21-item Depression, Anxiety, and Stress Scale (DASS-21) (DASS-21-Depression). A higher score indicates more anxiety symptoms with a minimum score of 0 and a maximum score of 21.
Stress levels at baseline in patients and family members | Baseline
  Stress as measured by the 7-item depression subscale of the self-reported 21-item Depression, Anxiety, and Stress Scale (DASS-21) (DASS-21-Depression). A higher score indicates more stress levels with a minimum score of 0 and a maximum score of 21.
Change in stress levels in patients and family members | Baseline + 30 days, baseline + 90 days, baseline + 180 days
  Stress as measured by the 7-item depression subscale of the self-reported 21-item Depression, Anxiety, and Stress Scale (DASS-21) (DASS-21-Depression). A higher score indicates more stress levels with a minimum score of 0 and a maximum score of 21.
Covid-19 related psychological stress at baseline in patients and family members | Baseline
  Specific distress regarding Covid-19 will be measured by the Dutch translation of the COVID-19 Peritraumatic Distress Index (CPDI). This self-reported questionnaire inquires about the frequency of anxiety, depression, specific phobias, cognitive change, avoidance and compulsive behaviour, physical symptoms and loss of social functioning in the past week. The score ranges from 0 to 100, with higher scores indicating more distress.
Change in Covid-19 related psychological stress in patients and family members | Baseline + 30 days, baseline + 90 days, baseline + 180 days
  Specific distress regarding Covid-19 will be measured by the Dutch translation of the COVID-19 Peritraumatic Distress Index (CPDI). This self-reported questionnaire inquires about the frequency of anxiety, depression, specific phobias, cognitive change, avoidance and compulsive behaviour, physical symptoms and loss of social functioning in the past week. The score ranges from 0 to 100, with higher scores indicating more distress.

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert MD Lemmens, MD, PhD, Study Director — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analyzed during the current study are not publicly available due to confidentiality issues but are available from the corresponding author upon reasonable request.